CLINICAL TRIAL: NCT04376034
Title: Convalescent Plasma Collection From Individuals That Recovered From COVID19 and Treatment of Critically Ill Individuals With Donor Convalescent Plasma
Brief Title: Convalescent Plasma Collection and Treatment in Pediatrics and Adults
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2004965705
Record Dates: First submitted 2020-04-19; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: COVID19; Coronavirus Infection; Coronavirus; Virus Diseases; RNA Virus Infections
Keywords: Covid19; Covid 19; Convalescent Plasma; SARS-CoV-2; Pediatric; Pediatrics
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases; RNA Virus Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild Severity (Other): Eligible to enroll in study and will be monitored for progression. Will not initially receive plasma.
  Interventions: Other: Standard of Care
- Moderate Severity (Active Comparator): Adult patients will be treated with 1 unit (200mL) of convalescent plasma
  Pediatric patients will be treated with 10mg/kg up to 1 unit of convalescent plasma.
  Interventions: Biological: Convalescent Plasma 1 Unit
- Severe or Critical Severity (Active Comparator): Adult patients will be treated with up to 2 units of convalescent plasma
  Pediatric patients will be treated with 10mg/kg up to 2 units of convalescent plasma.
  Interventions: Biological: Convalescent Plasma 2 Units

INTERVENTIONS:
Biological: Convalescent Plasma 1 Unit — Each adult recipient will receive 1 units of plasma, each unit will consist of about 200 to 250 mL.
  Each pediatric recipient will receive 10mL/kg up to 1 unit of plasma.
  Arms: Moderate Severity
Biological: Convalescent Plasma 2 Units — Those that meet severe or critical criteria will be given 2 units if available or 1 unit if 2 units are not available.
  Those that are given 1 unit may receive the second unit (or the remainder of the maximum pediatric weight calculated amount of plasma up to 1 additional unit) if they progress to severe or critical condition or if already in severe or critical condition but only received 1 unit secondary to shortages.
  Each pediatric recipient will receive 10mL/kg up to 2 units of plasma.
  Arms: Severe or Critical Severity
Other: Standard of Care — Those that meet mild severity will be allowed to enroll in the study, but will not receive plasma unless there is progression of illness into the moderate/rapid progression or greater category.
  Arms: Mild Severity

SUMMARY:
This is a prospective study, involving contacting potential plasma donors and the use of their plasma to help fight off infections of those suffering from COVID19 in accordance to collection guidelines for plasma and FDA IND requirement. This study will include up to 240 participants potentially receiving convalescent plasma and up to 1000 potential donors.

There are 3 basic arms to the study: mild, moderate and severe/critical severity. All 3 severity groups are eligible for enrollment, but mild severity will not be given plasma unless there is progression. Moderate severity will given up to 1 unit of plasma and severe/critical severity up to 2 units. There is no placebo group, however given the excepted issues of shortages of plasma, intention to treat will be used for analysis.

DETAILED DESCRIPTION:
Convalescent plasma (here on referred to as plasma) has been used in emergency life-threatening situations to treat infections for over 100 years. The plasma is donated by an individual that has recovered from the very same infection that another person is infected with. This plasma is enriched in the antibodies that recognize and helped the body's immune system fight off the infection. When transfused from donor to recipient those antibodies will aid the recipient in fighting off the infection. In recent history this has been used to fight Ebola. Recently, the Federal Food and Drug Agency (FDA) made possible expedited Investigational New Drug (IND) process for plasma use in the fight against COVID19 for emergency and lifesaving uses.

There are several other investigational drugs for treatment of COVID19 such as: Remdesivir, an antiviral. The off-label use of hydroxychloroquine, Lopinavir/ritonavir, or Tocilizumab have been authorized. Convalescent plasma mechanism of action helps to promote health by working with one's own immune system and will not interfere with the other proposed medications. It also will not weaken the immune system as the investigational and off label medications have the potential to do. Convalescent plasma is time honored and although investigational for each use against novel or rare infections, it is the basis for IgG infusions in the immunodeficient populations. Currently the use of IgG infusions such as Intravenous IgG (IVIG) is assumed to not have the right antibodies from donors in the general public. This is secondary to the novel nature of the COVID19 and the fact that the IVIG available today was collected 6 to 12 months ago from plasma donors; prior to the COVID19's outbreak discovery in China.

It is for that reason that IVIG is not recommended at this time and the FDA has made special fast-tracking announcements for plasma use for COVID19. Currently, plasma is the only treatment that has a previous history of success in these novel or rare viral outbreak situations. It has already been reported to have been associated with survival of 5 out of 5 participants in a pilot study in China

For the purpose of this study advanced respiratory support will include any measure of respiratory support above low flow nasal cannula oxygen (2 Liters/minute flow rate).

For the purpose of this study dyspnea will be defined as any shortness of breath that is not completely relieved with the use of low flow nasal canula oxygen set to 2 Liters/minute flow rate and/or requiring breathing treatments such as but not limited to: bronchodilators more than every 4 hours to relieve symptoms.

In the event that more than one recipient is identified and plasma is available in less than the total number of approved recipients, priority will be given to those approved by the FDA for the IND use of plasma for severe or critical condition. If there still exists a deficit of plasma, the priority will be given to those on advanced respiratory support with the most critical settings (if unclear then will be considered a tie); active pressor treatments; age <1 years of age with days of life, age adjusted for prematurity as a tie breaker; age >60 with years as a tie breaker; and lastly lottery pull with potential remaining recipients as the final tie breaker.

ELIGIBILITY:
Inclusion Criteria:

* Plasma donation:

  1. Prior diagnosis of COVID-19 documented by a laboratory test

     1. Abbott RealTime SARS-CoV-2 real-time reverse transcription polymerase chain reaction (rRT-PCR) test on the Abbott m2000 System (Inpatient WVU testing)
     2. Other testing methods and vendors using FDA approved detection methods of SARS-CoV-2 under the Emergency Use Authorization (EUA)
  2. Complete resolution of symptoms at least 28 days prior to donation
  3. Complete resolution of symptoms for at least 14 days with negative repeat COVID-19 testing approved by the FDA EUA
  4. Female donors age 18+ that have never been pregnant or negative for HLA antibodies
  5. Male donors age 18+
  6. Negative results for COVID-19 either from one or more nasopharyngeal swab specimens or by a molecular diagnostic test from blood. A partial list of available tests can be accessed at https://www.fda.gov/medical-devices/emergency-situations-medical-devices/emergency-use-authorizations.
  7. Defined SARS-CoV-2 neutralizing antibody titers, if testing can be conducted (e.g., of at least 1:1602, 1:360 up to 1:640 is preferred. In shortage case 1:80 is acceptable)
  8. At least or greater than 50kg of weight
* Plasma Recipients:

  1. Individuals of any age above 30 days of life, sex, or pregnancy status suffering from confirmed COVID19 and in rapid progression, severe or critical condition meeting the FDA IND guidelines.
  2. Must have laboratory confirmed COVID19
  3. Must have severe or immediately life-threatening COVID19
  4. Must provide informed consent/assent

Exclusion Criteria:

* Plasma donation:

  1. Individuals that do not meet the requirement from the American Red Cross for plasma donation or equivalent
  2. Individuals plasma that has not passed safety screening after procurement by the American Red Cross for plasma donation or equivalent
* Plasma Recipients

  1. Individuals with COVID19 who are not in clinical concern for rapid progression, severe or critical condition
  2. Individuals who are in critical condition that are not confirmed to have COVID19
  3. Individuals with known Selective IgA Deficiency, that has not been found to be absent of anti-IgA antibodies

Min Age: 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Donor | Measured in days for 365 days
  Time it takes to identify eligible donors whom are willing to donate
Plasma Donor | Measured in days for 365 days
  Time it takes the plasma collection center to contact willing donors whom are allowed to donate plasma
Plasma Recipient | Measured evey 24 hours up to 30 days
  Time from consent to infusion
Plasma Recipient | Measured in days with 30 day from discharge follow-up
  Survival

SECONDARY OUTCOMES:
Plasma Donor | Measured every 24 hours up to 1 year
  Time until plasma is donated
Plasma Recipient | Day 1, 2, 3, 4, 7, and 30 day
  Incident of treatment-Emergent Adverse Events [Safety and Tolerability]
Plasma Recipient | Day 1, 2, 3, 4, 7, and 30 day
  Morbidity reduction
Plasma Recipient | Measured every 24 hours until patient discharged from hospital up to 1 year
  Reduced Length of Stay in hospital
Plasma Recipient | Measured every 24 hours until Off Advanced Respiratory Support up to 1 year
  Reduced Length of Stay on Advance Respiratory Support

CONTACTS AND LOCATIONS:
Overall Officials: Brian Peppers, DO, PhD, Principal Investigator — WVU Medicine Children's
Locations (1):
- WVU Medicine, Morgantown, West Virginia, United States